CLINICAL TRIAL: NCT05693675
Title: Postoperative Oral Methadone After Major Spine Surgery; Safety, Feasibility and Efficacy in Prevention of Progression to Chronic Opioid Usage at 3 Months - A Pilot Trial.
Brief Title: Postoperative Oral Methadone After Major Spine Surgery; Safety, Feasibility and Efficacy in Prevention of Progression to Chronic Opioid Usage at 3 Months
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI left institution; no participants were enrolled
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Shobana Rajan, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-22-0912
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Spine Surgery
Keywords: opioids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Postoperative methadone (Experimental)
  Interventions: Drug: Postoperative methadone; Drug: Rescue Analgesia
- Postoperative placebo (Placebo Comparator)
  Interventions: Drug: Postoperative placebo; Drug: Rescue Analgesia

INTERVENTIONS:
Drug: Postoperative methadone — Participants will receive intraoperative methadone (0.2 mg/kg ideal body weight intravenously but not exceeding 20mg) followed by oral/IV methadone postoperatively according to the following scheme: A) Opioid naïve patients will receive 5mg twice daily dosage of methadone on postoperative days 1 and 2 followed by 5 mg daily on postoperative days 3, 4, and 5. B) Patients taking opioids preoperatively will continue to receive their regular opioids and additionally receive 5 mg twice a day of methadone on postoperative days 1 and 2, followed by 5 mg per day on days 3, 4 and 5.
  Arms: Postoperative methadone
Drug: Postoperative placebo — Participants will receive intraoperative methadone intravenously 0.2mg/kg followed by oral placebo postoperatively according to the following scheme: Opioid naïve patients and patients taking opioids preoperatively will receive placebo tablets twice daily on day 1 and day 2 and once daily day 3, 4 and 5. Patients taking preoperative opioids will be able to return to their baseline opioids immediately after surgery.
  Arms: Postoperative placebo
Drug: Rescue Analgesia — PACU analgesia for both groups will be the usual care regime of fentanyl or hydromorphone bolus as prescribed by the physician anesthesiologist doing the case. All patients receive IV intravenous patient-controlled analgesia and rescue opioids which is usual care for postoperative pain.

SUMMARY:
The purpose of this study is to evaluate the feasibility and safety of a clinical protocol based on the administration of intraoperative intravenous methadone followed by a short regimen of oral/IV (if the patient is not able to take oral) methadone following spine surgery and to evaluate if methadone decreases persistent opioid usage at 3 months in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing multilevel complex lumbar and/or thoracic spine fusion surgery, including revision surgeries

Exclusion Criteria:

* BMI greater than 40

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of study design as assessed by the number of participants for which scheduled postoperative methadone versus placebo were able to be administered according to the scheme described | Day of discharge (about 6 days after surgery)
Feasibility of study design as assessed by number of participants for which safety was able to be assessed (EKGs) | postop days 1 and 5
Feasibility of study design as assessed by the number of participants for which safety was able to be assessed (respiratory events) | Day of discharge (about 6 days after surgery)
  ability to evaluate adverse respiratory events
Feasibility of study design as assessed by the number of participants for which postop opioid usage could be surveyed at 3 months | 3 months after surgery

SECONDARY OUTCOMES:
Number of participants for which opioid usage was able to be collected | Day of discharge (about 6 days after surgery)
Safety as assessed by the number of patients developing respiratory depression | by fifth day of hospital stay
  Saturation of Oxygen(SPO2) less than 85%, Respiratory rate <5 for longer than 3 minutes, ( Khanna et) increased oxygen requirement related to opioid-induced respiratory depression, naloxone use. The SPO2 will be monitored continuously per usual care in post anesthesia care unit (PACU) and every 4 hours in the ward.
Safety as assessed by the number of patients developing clinically significant corrected QT interval(QTc )prolongation | by fifth day of hospital stay
  QTc interval >500ms or >25% increase from baseline; number of patients developing arrhythmias needed treatment
Safety as assessed by the number of participants with hallucinations | by fifth day of hospital stay
Safety as assessed by the number of participants with dizziness | by fifth day of hospital stay
Safety as assessed by the number of participants with Antiemetic use | by fifth day of hospital stay
Safety as assessed by the number of participants with occurrence of nausea | by fifth day of hospital stay
Safety as assessed by the number of participants with occurrence of vomiting | by fifth day of hospital stay
Safety as assessed by the number of participants with occurrence of Ileus or constipation | by fifth day of hospital stay
Safety as assessed by the number of subjects with persistent opioid use | 3 months after surgery
  This is scored from 0(less than once a week) to 4(constantly, a higher number indicating more opioid use)

CONTACTS AND LOCATIONS:
Overall Officials: Shobana Rajan, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No